CLINICAL TRIAL: NCT03000127
Title: A Pilot Trial of Testosterone Treatment for Fatigue in Men With Multiple Sclerosis
Brief Title: Testosterone for Fatigue in Men With MS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of California, Los Angeles (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Rhonda Voskuhl, Professor, Department of Neurology, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01NS102295
Record Dates: First submitted 2016-12-17; First posted 2016-12-21 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis
Keywords: testosterone; multiple sclerosis; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Testosterone; Gels

STUDY DESIGN:
Intervention Model Description: Single arm, testosterone or placebo will be administered to all patients at some period of study, but which period of study the they will recieve placebo or testosterone gel will be blinded (unknown) to participant, care provider, and outcomes assessor.
Masking Description: All patients will receive either testosterone or placebo at some phase of treatment, but which phase will be testosterone and which will be placebo will be unknown (blinded) to participant, care provider, and outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm crossover (Experimental): All patients will receive testosterone gel and placebo gel during some months, but the months that they are on each treatment will be unknown to the patient
  Interventions: Drug: AndroGel 1 % Topical Gel; Drug: Placebos

INTERVENTIONS:
Drug: AndroGel 1 % Topical Gel — testosterone gel
Drug: Placebos — Placebo gel

SUMMARY:
Fatigue is a major symptom in people with multiple sclerosis (MS), for which treatments are limited. Several studies have shown that a large proportion of men with MS have low testosterone levels. We propose a two-site clinical trial using topical testosterone gel as a treatment for MS-related fatigue in men with progressive MS who have low or low-normal testosterone levels.

ELIGIBILITY:
Inclusion Criteria:

1) Men with SPMS or PPMS, 2)18-60 years old, 3) EDSS of 1.0- 6.5, 4) Low or low-normal T < 499ng/dL and 5) FSS scores of >3.6.

Exclusion Criteria:

1) Prostate specific antigen > 2.5 (<49yr of age) or >3.5 (age >50yr of age), 2) baseline hematocrit greater than the upper limit of normal for the laboratory used, 3) EKG with ischemic changes, 4) history of myocardial infarction, unstable angina, stroke, transient ischemic attack, or deep vein thrombosis, 5) history of prostate or breast cancer, 6) screening T level >500ng/dL, 7) diabetes requiring treatment, 8) current drug/alcohol abuse, 9) disease other than MS causing fatigue, such as obstructive sleep apnea or other sleep disorder, or untreated thyroid dysfunction, 10) RRMS, 11) Beck Depression Inventory-II (BDI) score over 20, 12) cognitive dysfunction such that subject cannot perform study tests, 13) inability to undergo MRI, 14) current or expected use of amphetamines, or 15) anticipated changes in medical treatments that might affect fatigue scores (e.g., expected changes in spasticity, sleep, or depression medications).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | 18 months
  assessment of fatigue severity

SECONDARY OUTCOMES:
Localized Gray Matter Atrophy | 18 months
  Quantify effect of testosterone treatment on localized gray matter atrophy
Axon Density in White Matter | 18 months
  Quantify effect of testosterone treatment on axon density in major white matter tracts

OTHER OUTCOMES:
Correlation of testosterone level with fatigue | 18 months
Correlation of localized gray matter atrophy with fatigue | 18 months
Correlation of axon density in white matter with fatigue | 18 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sicotte NL, Giesser BS, Tandon V, Klutch R, Steiner B, Drain AE, Shattuck DW, Hull L, Wang HJ, Elashoff RM, Swerdloff RS, Voskuhl RR. Testosterone treatment in multiple sclerosis: a pilot study. Arch Neurol. 2007 May;64(5):683-8. doi: 10.1001/archneur.64.5.683. PMID 17502467
- [Background] Kurth F, Luders E, Sicotte NL, Gaser C, Giesser BS, Swerdloff RS, Montag MJ, Voskuhl RR, Mackenzie-Graham A. Neuroprotective effects of testosterone treatment in men with multiple sclerosis. Neuroimage Clin. 2014 Mar 6;4:454-60. doi: 10.1016/j.nicl.2014.03.001. eCollection 2014. PMID 24634831
- [Background] Gold SM, Chalifoux S, Giesser BS, Voskuhl RR. Immune modulation and increased neurotrophic factor production in multiple sclerosis patients treated with testosterone. J Neuroinflammation. 2008 Jul 31;5:32. doi: 10.1186/1742-2094-5-32. PMID 18671877
- [Background] Ziehn MO, Avedisian AA, Dervin SM, Umeda EA, O'Dell TJ, Voskuhl RR. Therapeutic testosterone administration preserves excitatory synaptic transmission in the hippocampus during autoimmune demyelinating disease. J Neurosci. 2012 Sep 5;32(36):12312-24. doi: 10.1523/JNEUROSCI.2796-12.2012. PMID 22956822
- [Background] Gold SM, Voskuhl RR. Estrogen and testosterone therapies in multiple sclerosis. Prog Brain Res. 2009;175:239-51. doi: 10.1016/S0079-6123(09)17516-7. PMID 19660660
- [Background] Liva SM, Voskuhl RR. Testosterone acts directly on CD4+ T lymphocytes to increase IL-10 production. J Immunol. 2001 Aug 15;167(4):2060-7. doi: 10.4049/jimmunol.167.4.2060. PMID 11489988
- [Background] Dalal M, Kim S, Voskuhl RR. Testosterone therapy ameliorates experimental autoimmune encephalomyelitis and induces a T helper 2 bias in the autoantigen-specific T lymphocyte response. J Immunol. 1997 Jul 1;159(1):3-6. PMID 9200430
- [Background] Golden LC, Voskuhl R. The importance of studying sex differences in disease: The example of multiple sclerosis. J Neurosci Res. 2017 Jan 2;95(1-2):633-643. doi: 10.1002/jnr.23955. PMID 27870415
- [Background] Spence RD, Voskuhl RR. Neuroprotective effects of estrogens and androgens in CNS inflammation and neurodegeneration. Front Neuroendocrinol. 2012 Jan;33(1):105-15. doi: 10.1016/j.yfrne.2011.12.001. Epub 2011 Dec 24. PMID 22209870
- [Background] Hussain R, Ghoumari AM, Bielecki B, Steibel J, Boehm N, Liere P, Macklin WB, Kumar N, Habert R, Mhaouty-Kodja S, Tronche F, Sitruk-Ware R, Schumacher M, Ghandour MS. The neural androgen receptor: a therapeutic target for myelin repair in chronic demyelination. Brain. 2013 Jan;136(Pt 1):132-46. doi: 10.1093/brain/aws284. PMID 23365095
- [Background] Voskuhl RR, Gold SM. Sex-related factors in multiple sclerosis susceptibility and progression. Nat Rev Neurol. 2012 Mar 27;8(5):255-63. doi: 10.1038/nrneurol.2012.43. PMID 22450508